CLINICAL TRIAL: NCT05956106
Title: Therapeutic Effect of Mulberry Fruit Powder Consumption in Metabolic Syndrome
Brief Title: Effect of Mulberry Fruit Powder in Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Asif Ali, Lecturer, Department of Food Sciences and Human Nutrition, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Mulberry Fruit Powder
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Syndrome
Keywords: Hypertension; Diabetes; Obesity; Hyperlipidemia; Mulberry; Anthocyanin
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Diabetes Mellitus; Obesity; Hyperlipidemias | interventions — morniga G protein, Morus nigra

STUDY DESIGN:
Intervention Model Description: Case-Control Study
Masking Description: Participants groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic syndrome patients (Experimental): Dried Mulberry fruit powder is used for preventing symptoms in Metabolic Syndrome patients Dietary intervention: Black Mulberry fruit powder Dosage: 45g per day
  Interventions: Dietary Supplement: Black Mulberry Fruit Powder

INTERVENTIONS:
Dietary Supplement: Black Mulberry Fruit Powder — Anthocyanin plays a major role in preventing symptoms of metabolic syndrome.
  Other Names: Morus Nigra

SUMMARY:
Metabolic syndrome is a raising concern globally, especially in developing countries such as Pakistan. To prevent its risk factors diet and lifestyle modification is major solution. Functional foods have additional benefits of treating disease while providing basic nutrients. Mulberry is a native fruit with the properties of functional food, it is rich in anthocyanin and different anti-obesity,anti-diabetic, and anti-hyperlipidemic treating potential antioxidants. Mulberry will prove its therapeutic potential against the risk factors of metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic syndrome, which is characterized by a number of concurrent risk factors. These risk factors include dysglycemia, high blood pressure, high triglyceride levels, low levels of HDL cholesterol, and obesity (particularly central adiposity). It is rapidly increasing the burden of non-communicable diseases (NCDs) in Pakistan. The prevalence of MetS in Pakistan is 28.6%, and suburban areas from the province of Punjab showed a high prevalence. Females are more prone to metabolic syndrome. Dietary and lifestyle modification can prevent MetS from converting into CVD, T2DM, and stroke. There is limited documented research in Pakistan related to the therapeutic roles of mulberry fruit powder. With respect to these limitations, the present study aims to assess the therapeutic roles of mulberry fruit powder consumption on metabolic syndrome.

The utilization of dried mulberry fruit powder (MFP) as a component of nutritional supplementation will effectively ameliorate the clinical markers associated with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having fasting total cholesterol level of ≥ 200 mg/dl or LDL cholesterol ≥ 130 mg/dl.
* Fasting Blood Glucose ≥110mg/dl.
* SBP ≥ 130/ ≥ 85 mmHg
* Waist Circumference of ≥40 inches in males and ≥35 inches for females

Exclusion Criteria:

* Participants of age 55 or above
* Participants who have less than two risk factors

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Lipid profile will be assessed before and after the trial. | 45 days
  The change in lipid profile, after consuming mulberry fruit powder for 45 days, will be assessed. The value will be closed to optimized values.
Fasting glucose level will be assessed before and after the trial | 45 days
  The change in fasting glucose levels will be assessed after consuming mulberry fruit powder for 45 days.The values will be become close to optimized levels
Weight circumference will be measured before and after the trial | 45 days
  The change in weight will be measured after consuming mulberry fruit powder for 45 days.The value will be close to normal range.
Blood pressure will be assessed before and after the trial. | 45 days
  The change in systolic and diastolic blood pressure, after consuming mulberry fruit powder for 45 days. The values will become close to optimized levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Shan Medicare Hospital, Arifwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
All available data will be confidential

REFERENCES:
- [Result] Wan M, Li Q, Lei Q, Zhou D, Wang S. Polyphenols and Polysaccharides from Morus alba L. Fruit Attenuate High-Fat Diet-Induced Metabolic Syndrome Modifying the Gut Microbiota and Metabolite Profile. Foods. 2022 Jun 20;11(12):1818. doi: 10.3390/foods11121818. PMID 35742014
- See also: Polyphenols and Polysaccharides from Morus alba L. Fruit Attenuate High-Fat Diet-Induced Metabolic Syndrome — https://pubmed.ncbi.nlm.nih.gov/35742014/